CLINICAL TRIAL: NCT04469634
Title: Are SARS-CoV-2 Specific Antibodies a Correlate for Protection?
Acronym: ImmCoV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Jessa Hospital (Other); University Hospital, Antwerp (Other); Universiteit Antwerpen (Other); Sciensano (Other Government); Mensura (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1412/20
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- antibody response and memory B-cell (Experimental): Regular blood draws to measure antibody responses and memory B-cell responses Regular swab collection to test for re-infection
  Interventions: Diagnostic Test: Assessing antibody responses, neutralizing capacity and memory B-cell function

INTERVENTIONS:
Diagnostic Test: Assessing antibody responses, neutralizing capacity and memory B-cell function — Assessing antibody responses, neutralizing capacity and memory B-cell function and their contribution to protection against re-infection

SUMMARY:
The objectives of this study are (1) to determine the ex vivo neutralizing capacity and the longevity of SARS-CoV-2-specific Ab responses and (2) to measure the memory B-cell responses in a cohort of health care workers (HCW) recovering from severe, mild or asymptomatic infection. By focusing on HCW, a population that is at risk for re-infection during a second epidemic wave, the correlation between nAb levels and protection is investigated.

DETAILED DESCRIPTION:
SARS-CoV-2 has spread at an unprecedented speed and scale since January 2020. Since then, Belgium has been confronted with >60.000 diagnosed cases and likely many more undiagnosed with mild or no symptoms. The true seroprevalence of SARS-CoV-2 in the Belgian population is not known, yet increasing confidence about the performance of several serological assays paves the way to large-scale serosurveys. These studies will be crucial in assessing population immunity and evaluating the risk of re-infection. The first, smaller-scaled, antibody surveys report a range of seroprevalences, i.e. Germany (14%), The Netherlands (4%), USA (2.49-4.16%) and Belgium (4.7-6.9%). These studies suffer from conceptual and technical flaws yet are used for easing lockdown measures. A major limitation is that antibody (Ab) capture assays measure exposure to SARS-CoV-2, rather than subsequent protection, which requires assessment of the quality of the Abs including their capacity to neutralize the virus. Also the Ab levels required for protection and their duration are yet unknown. The proposed project aims to address these pertinent questions in a population at risk of re-infection during a second epidemic wave. Sero-neutralisation assays are regarded the gold standard method to measure ex vivo Ab neutralising activity against viruses, including SARS-CoV-2. A recent Chinese study, using a pseudovirus neutralisation assay, found that nAbs are detected from day 10-15 after onset of disease and that younger patients typically have lower levels of nAbs compared to middle-aged and elderly patients. Importantly, in about 1 out of 3 patients the nAb titers were low and in 10 young patients nAbs were absent. A pseudovirus is an imperfect model for SARS-CoV-2 because of the non-natural embedding of Spike protein in the pseudovirions and differences in glycosylation. In this study, a whole virus neutralisation assay will be used that was recently validated using a panel of SARS-CoV-2 convalescent sera in the lab of the Principal Investigator. Preliminary results of the study team show a rapid decline in nAb titer within 15-36d after diagnosis in 4/11 patients, while IgG and IgA remain steady and high in ELISA. Older studies with SARS-CoV-1 showed declining IgM and IgA antibody titers within 6 months, declining IgG titers after 1y, and a complete lack of antigen-specific peripheral memory B-cell (MBC) responses after recovery. Measuring only circulating Abs can be misleading as it excludes the detection of the MBC pool, which can exist in the absence of detectable serum Ab levels and is a pre-requisite to maintain protective immunity in the long term. Upon re-encounter with the antigen, MBC can rapidly differentiate to produce Abs. So far, little is known about humoral immune responses against SARS-CoV-2 and their contribution to protection.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed (PCR+) with COVID-19 between March-May 2020
* Be a permanent employee (HCW: nurse, physician, paramedical) of the study hospital
* Agree to complete a short questionnaire and be sampled 4 tubes of heparin whole blood every 3 months over a one-year period
* Have given their informed consent to participate

Exclusion Criteria:

* Persons in serious clinical condition, incompatible with the informed consent procedure
* Pregnant women
* Persons that have not been diagnosed with COVID-19

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Antibody levels over time | 12 months
  Antibody levels over time
Antibody neutralizing capacity | 12 months
  Antibody neutralizing capacity
Memory B-cell function | 12 months
  Memory B-cell function
Antibody-dependent enhancement | 12 months
  Antibody-dependent enhancement

SECONDARY OUTCOMES:
Re-infection with SARS-CoV2 | 12 months
  Re-infection with SARS-CoV2

CONTACTS AND LOCATIONS:
Overall Officials: Kevin K. Ariën, PhD, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - Jessa Hospital, Hasselt

IPD SHARING:
Plan to Share IPD: Undecided